CLINICAL TRIAL: NCT00003222
Title: Phase II Trial for the Evaluation of the Efficacy of Vaccination With Synthetic Melanoma Peptides Either Pulsed on Dendritic Cells, or Administered With GM-CSF-in-Adjuvant, Plus Administration of Sustemic IL-2, in Patients With Advanced Melanoma.
Brief Title: Vaccine Therapy Plus Interleukin-2 in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Craig L Slingluff, Jr, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7621; IRB-HSR 7621; NCI-G98-1389
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2; incomplete Freund's adjuvant; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peptides pulsed on dendritic cells (Experimental): 4 melanoma peptides pulsed on monocyte-derived dendritic cells
  Interventions: Biological: aldesleukin; Biological: gp100 antigen; Biological: incomplete Freund's adjuvant; Biological: tetanus peptide melanoma vaccine; Biological: tyrosinase peptide
- Peptides in GMCSF-in-adjuvant (Experimental): 4 melanoma peptides administered as an emulsion with GM-CSF and Montanide ISA-51 adjuvant.
  Interventions: Biological: aldesleukin; Biological: gp100 antigen; Biological: incomplete Freund's adjuvant; Biological: sargramostim; Biological: tetanus peptide melanoma vaccine; Biological: tyrosinase peptide

INTERVENTIONS:
Biological: aldesleukin — Systemic subcutaneous delivery of low-dose IL-2.
  Other Names: Interleukin-2
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: sargramostim
  Arms: Peptides in GMCSF-in-adjuvant
Biological: tetanus peptide melanoma vaccine
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines made from melanoma cells may make the body build an immune response to and kill tumor cells. Colony-stimulating factors such as GM-CSF may increase the number of immune cells found in the bone marrow or peripheral blood. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells. Combining vaccine therapy with GM-CSF and interleukin-2 may be kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccines made from melanoma cells with or without GM-CSF followed by interleukin-2 in treating patients with stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effectiveness of vaccination with synthetic melanoma peptides pulsed on autologous dendritic cells versus vaccination with synthetic melanoma peptides plus sargramostim (GM-CSF) in decreasing tumor burden in patients with high risk melanoma (pulsed autologous dendritic cell arm closed 1/8/2001). II. Determine whether these regimens result in increased tumor specific immune responses as measured in vitro and in vivo. III. Determine whether these regimens stimulate T-cell responses in these patients.

OUTLINE: This is an open label study. Patients are included in treatment arm II only (arm I closed 1/8/2001): Arm I: Patients undergo leukapheresis to collect dendritic cells. Patients receive a mixture of synthetic melanoma peptides (gp100 antigen, tyrosinase, and tetanus peptides) pulsed on autologous dendritic cells IV and subcutaneously (SC). Arm II: Patients receive a mixture of synthetic melanoma peptides (gp100 antigen, tyrosinase, and tetanus peptides) and sargramostim (GM-CSF) emulsified in Montanide ISA-51 SC and intradermally. Patients receive vaccination during weeks 0, 1, 2, 4, 5, and 6 for a total of 6 doses and interleukin-2 SC daily on days 7-49. Patients receive 3 additional vaccinations at different sites not involved with the tumor concurrently with the first 3 vaccinations. Patients are evaluated at 8 weeks, 12 weeks, 6 months, 12 months, and 24 months.

PROJECTED ACCRUAL: A total of 27-54 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage III or IV melanoma gp100 positive tumor cells and/or tyrosinase positive tumor cells HLA type A1, A2, or A3 Measurable disease May have up to 3 brain metastases if all are less than 2 cm in diameter and are asymptomatic, and there is no mass effect or they have been treated successfully by surgical excision or by gamma knife radiation therapy

PATIENT CHARACTERISTICS: Age: 18 to 79 Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: Bilirubin no greater than 2.5 times upper limit of normal (ULN) AST and ALT no greater than 2.5 times ULN Alkaline phosphatase no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No New York Heart Association class II, III, or IV heart disease Other: No known or suspected allergy to any component of the vaccine No medical condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 months since prior growth factors At least 3 months since prior agents with putative immunomodulating activity (except nonsteroidal antiinflammatory agents) At least 1 year since other prior melanoma vaccinations Chemotherapy: At least 3 months since prior chemotherapy No concurrent chemotherapy Endocrine therapy: At least 3 months since prior corticosteroids No concurrent corticosteroids Radiotherapy: At least 3 months since prior radiotherapy No concurrent radiotherapy Surgery: See Disease Characteristics Other: At least 3 months since other prior investigational drugs or therapy At least 3 months since prior allergy desensitization injections At least 14 days since completion of acute treatment for a serious infection No concurrent allergy desensitization injections

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-04; Primary Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, MD, Study Chair — University of Virginia
Locations (1):
- Cancer Center at the University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Slingluff CL Jr, Petroni GR, Yamshchikov GV, Barnd DL, Eastham S, Galavotti H, Patterson JW, Deacon DH, Hibbitts S, Teates D, Neese PY, Grosh WW, Chianese-Bullock KA, Woodson EM, Wiernasz CJ, Merrill P, Gibson J, Ross M, Engelhard VH. Clinical and immunologic results of a randomized phase II trial of vaccination using four melanoma peptides either administered in granulocyte-macrophage colony-stimulating factor in adjuvant or pulsed on dendritic cells. J Clin Oncol. 2003 Nov 1;21(21):4016-26. doi: 10.1200/JCO.2003.10.005. PMID 14581425

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 participants were assigned to each arm in Stage I. 14 additional participants were assigned in Stage II to study arm 2. Data are reported for stage I. Reporting is planned for stage II when data are available.
Groups:
- Peptides Pulsed on Dendritic Cells: ---peptides were pulsed on monocyte-derived dendritic cells cultures in GM-CSF and IL-4
- Peptides in Sargramostim (GMCSF)-In-Montanide ISA-51 Adjuvant: ---Peptides were administered in an emulsion of sargramostim (GM-CSF) and Montanide ISA-51 (incomplete Freund's) adjuvant
Period: Overall Study
Arm/Group | Peptides Pulsed on Dendritic Cells | Peptides in Sargramostim (GMCSF)-In-Montanide ISA-51 Adjuvant
Started | 13 | 28
Completed | 13 | 27 (Decline in performance status between enrollment and initiation of therapy.)
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peptides Pulsed on Dendritic Cells | Peptides in GMCSF-in-adjuvant | Total
Number analyzed (Participants) | 13 | 28 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 23 | 32
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13) | 55 (11) | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 6 | 19 | 25
Region of Enrollment [Number; unit: participants]
  United States | 13 | 28 | 41

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Objective Clinical Response (CR/PR/SD)
Description: The primary end point for this trial was clinical response. This was assessed by measurement of assessable metastatic deposits by CT, MRI, or direct measure of cutaneous deposits. Baseline tumor measurements used for assessment of clinical response were those obtained most immediately before the first vaccine administration and within 6 weeks of protocol entry. Measurements were made and reviewed by a multidisciplinary team. The original protocol defined tumor response on the basis of changes in cross-sectional area calculated as the product of two perpendicular measures. However, since the initiation of this study, the Response Evaluation Criteria in Solid Tumors Group (RECIST) system was employed as the current standard for clinical trials, in which response is based on changes in maximum cross-sectional dimensions. Computed tomography scans of clinical responders were reviewed again by a senior faculty radiologist not otherwise involved in the study.
Time Frame: Weeks 0-6,12; Months 6,12 and 24
Population: The analysis of this outcome measure was performed on subjects enrolled in Stage I of the trial, which included 13 subjects in each arm.
Measure: Number; unit: participants
Arm/Group | Peptides Pulsed on Dendritic Cells | Peptides in GMCSF-in-adjuvant
Number analyzed (Participants) | 13 | 13
participants
  Complete Response | 0 | 0
  Partial Response | 1 | 2
  Stable Disease | 1 | 2
  Progressive Disease | 11 | 9

2. Primary Outcome: Measure of Tumor-antigen-specific Immunity in Peripheral Blood Mononuclear Cells (PBMC) by Elispot Assay
Time Frame: Weeks 0-6,12; Months 6,12 and 24
Population: The analysis of this outcome measure was performed on subjects enrolled in Stage I of the trial, which included 13 subjects in each arm. Some patients were not evaluable because of inadequate sample availability.
Measure: Number; unit: responders
Arm/Group | Peptides Pulsed on Dendritic Cells | Peptides in GMCSF-in-adjuvant
Number analyzed (Participants) | 9 | 12
responders | 1 | 5
Statistical Analysis 1: Comparison: Peptides Pulsed on Dendritic Cells vs Peptides in GMCSF-in-adjuvant; This is a test for differences between the response rates of the two arms. The null hypothesis is that the arms have equal response rates and the alternative hypothesis is that they are different; Test type: Superiority or Other; p = 0.13, Chi-squared

3. Primary Outcome: Measure of Tumor-antigen-specific Immunity in Sentinel Immunized Node (SIN) by Elispot Assay
Time Frame: Weeks 0-6,12; Months 6,12 and 24
Population: Analysis of this outcome measure was performed on subjects in Stage I of the trial. Sentinel immunized nodes (SIN) were not evaluable for early tumor progression (5 arm 1, 2 arm 2) and patient refusal (1 arm 2). Thus, SINs were evaluable from 8 in arm 1 and 10 on arm 2, exceeding the protocol requirement for at least 6 subjects on each arm.
Measure: Number; unit: responders
Arm/Group | Peptides Pulsed on Dendritic Cells | Peptides in GMCSF-in-adjuvant
Number analyzed (Participants) | 8 | 10
responders | 1 | 8
Statistical Analysis 1: Comparison: Peptides Pulsed on Dendritic Cells vs Peptides in GMCSF-in-adjuvant; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.004, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 years
Description: Toxicity was recorded with a daily diary of toxicities, reviewed by the research team and supplemented by direct questioning, for the as treated population. Among patients assigned to arm 1, 3 patients progressed rapidly during DC preparation and required other interventions that caused removal from this study before the first vaccine.
Arm/Group | Peptides Pulsed on Dendritic Cells | Peptides in GMCSF-in-adjuvant
Serious Adverse Events (participants affected / at risk) | 0/10 | 5/27
Other Adverse Events (participants affected / at risk) | 9/10 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peptides Pulsed on Dendritic Cells (N=10) | Peptides in GMCSF-in-adjuvant (N=27)
Alkaline Phosphatase (Hepatobiliary disorders) | 0 | 1
Creatinine (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Fever (General disorders) | 0 | 1
General- Other (Cardiac disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Nervous system disorders) | 0 | 1
Other (Endocrine disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peptides Pulsed on Dendritic Cells (N=10) | Peptides in GMCSF-in-adjuvant (N=27)
Alkaline Phosphatase (Hepatobiliary disorders) | 0 | 8
Anorexia (Gastrointestinal disorders) | 4 | 17
Arthralgia (General disorders) | 0 | 2
Bilirubin (Hepatobiliary disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Diarrhea (Gastrointestinal disorders) | 4 | 10
Dizziness/Lightheadedness (Nervous system disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Edema (Cardiac disorders) | 1 | 6
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Fatigue (General disorders) | 8 | 26
Fever (General disorders) | 4 | 17
Flushing (Skin and subcutaneous tissue disorders) | 2 | 6
Headache (General disorders) | 4 | 17
Hemoglobin (Blood and lymphatic system disorders) | 1 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 7
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 4
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 6 | 24
Insomnia (Nervous system disorders) | 0 | 2
Mood (Nervous system disorders) | 1 | 4
Myalgia (General disorders) | 0 | 4
Myalgia/Arthralgia (General disorders) | 3 | 14
Nausea (Gastrointestinal disorders) | 5 | 17
Other (Eye disorders) | 0 | 2
Other (General disorders) | 1 | 1
Other PAIN (General disorders) | 2 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 14
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 0 | 4
Rigors, Chills (General disorders) | 5 | 20
SGOT (AST) (Hepatobiliary disorders) | 0 | 2
SGOT/SGPT (Hepatobiliary disorders) | 1 | 3
SGPT (ALT) (Hepatobiliary disorders) | 0 | 5
Skin (Skin and subcutaneous tissue disorders) | 1 | 3
Skin Rash/Urticaria (Skin and subcutaneous tissue disorders) | 4 | 4
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 1 | 5
Sweating (General disorders) | 3 | 11
Voice Changes/Stridor/Larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 2 | 6
Weight Gain/Loss (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes